CLINICAL TRIAL: NCT00233441
Title: Placebo Controlled Double Blind Dose Ranging Study of the Efficacy and Safety of SSR149744C 50, 100, 200, or 300 mg OD, With Amiodarone as Calibrator for the Maintenance of Sinus Rhythm in Patients With Recent Atrial Fibrillation/Flutter
Brief Title: Placebo Controlled Double-blind Dose Ranging Study of the Efficacy and Safety of SSR149744C 50, 100, 200 or 300 mg OD With Amiodarone as Calibrator for the Maintenance of Sinus Rhythm in Patients With Recent Atrial Fibrillation/Flutter
Acronym: MAIA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5165
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Arrhythmia; Anti-Arrhythmia Agents
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac | interventions — celivarone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: CELIVARONE (SSR149744C)

SUMMARY:
Double blind study to evaluate the efficacy and tolerability of SSR149744C and select a dose to be further investigated in the maintenance of sinus rhythm after electrical, pharmacological or spontaneous conversion of AF/AFL.

DETAILED DESCRIPTION:
This is a dose-ranging multicenter, multinational, randomized, double-blind, placebo-controlled, parallel arm study with 4 SSR149744C dose regimens and amiodarone as a calibrator.To be eligible, patients must be in normal sinus rhythm for at least one hour at randomization and must have an electrocardiogram documented history of recent AF/AFL reverted to normal sinus rhythm by electrical, pharmacological or spontaneous conversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years or more of either sex with documented sinus rhythm for at least 1 hour at the time of randomization with at least one ECG-documented AF/AFL episode in the last 3 months.

Exclusion Criteria:

* MAIN CRITERIA (non-exhaustive list):Women of childbearing potential without adequate birthcontrol, Pregnant Women, Breastfeeding women, contraindications to amiodarone, conditions which increase the risk of severe antiarrhythmic drug side effects, severe left ventricular dysfunction, severe associated conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the time from randomization to first documented AF/AFL recurrence indicated by 12-lead ECG or trans-telephonic ECG monitoring tracings showing AF/AFL.

SECONDARY OUTCOMES:
The secondary endpoints will be the following:time from randomization to first symptomatic AF/AFL recurrence - mean ventricular rate during AF/AFL at first recorded AF/AFL recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (17):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Tokyo, Japan
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Result] Khitri AR, Aliot EM, Capucci A, Connolly SJ, Crijns H, Hohnloser SH, Kulakowski P, Roy D, Radzik D, Kowey PR. Celivarone for maintenance of sinus rhythm and conversion of atrial fibrillation/flutter. J Cardiovasc Electrophysiol. 2012 May;23(5):462-72. doi: 10.1111/j.1540-8167.2011.02234.x. Epub 2011 Dec 15. PMID 22171925